CLINICAL TRIAL: NCT06743035
Title: Ropeginterferon Alfa-2b in Patients With Polycythemia Vera (PV) Without Symptomatic Splenomegaly: A Prospective, Longitudinal, Multicenter, Observational Study in Germany
Brief Title: Ropeginterferon Alfa-2b in Patients With Polycythemia Vera (PV) Without Symptomatic Splenomegaly
Acronym: ROPE
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: AOP Orphan Pharmaceuticals Germany GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOM-060513
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Polycythemia Vera
Keywords: Ropeginterferon alfa-2b; polycythemia vera; symptom burden; myeloproliferative neoplasm
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this non interventional study is to evaluate symptom burden in adult patients with PV without symptomatic splenomegaly during treatment with ropeginterferon alfa-2b in a real-world setting. Further patient-relevant endpoints include effectiveness including complete hematologic response (CHR), event-free survival (EFS), safety and tolerability, treatment reality including dosing details as well as factors affecting treatment decision making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed diagnosis of PV without symptomatic splenomegaly
* Indication and decision for treatment with ropeginterferon alfa-2b in accordance with current SmPC
* No prior treatment with ropeginterferon alfa-2b (Patients are allowed to be enrolled up to 6 weeks after their first dose of ropeginterferon alfa-2b but must still be on treatment at the time of enrollment.)
* Dated signature of informed consent form
* Participation in Patient-Reported Outcome (PRO) assessment in German language and completion of questionnaire at time of study enrollment
* Other criteria according to current Summary of Product Characteristics

Exclusion Criteria:

* Participation in an interventional clinical trial (except follow-up)
* Other contraindications according to current Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with polycythemia vera (PV) without symptomatic splenomegaly with the decision for treatment with ropeginterferon alfa 2b according to Summary of Product Characteristics (SmPC).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Symptom Burden | From Time of enrollment until month 36.
  Absolute values of the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) total symptom score (TSS) at time of study enrollment, during course of study until month 36.

SECONDARY OUTCOMES:
Effectiveness: Complete hematologic response (CHR) rate | From time of treatment start until end of study (max. 54 months after FPI)
  CHR rate is defined as the proportion of patients with
  * Hematocrit (HCT) <45% and
  * Phlebotomy-free (absence of phlebotomy during the previous 3 months) and
  * Platelet count ≤400 x 10^9/L and
  * white blood cell count ≤10 x 10^9/L
Effectiveness: Event-free survival (EFS) | From time of treatment start until end of study (max. 54 months after FPI)
  EFS is defined as the time from the first administration of ropeginterferon alfa-2b until the first occurrence of a thromboembolic event, disease progression to post-PV myelofibrosis, acute myeloid leukemia (AML) transformation, or death, whichever comes first. Patients without any event at the time point of analysis will be censored with their respective date of last contact.
Effectiveness: Proportion of patients with platelet count ≤400 ×109/L | From time of treatment start until end of study (max. 54 months after FPI)
  Platelet count (descriptive statistics and frequencies ≤400 vs. > 400 ×109/L)
Effectiveness: Proportion of patients with WBC count <10 ×109/L | From time of treatment start until end of study (max. 54 months after FPI)
  WBC count (descriptive statistics and frequencies <10 vs. ≥10 ×109/L)
Effectiveness: Proportion of patients with HCT value <45% | From time of treatment start until end of study (max. 54 months after FPI)
  HCT value (descriptive statistics and frequencies <45% vs. ≥45%)
Effectiveness: Proportion of patients without phlebotomy during course of study | From time of treatment start until end of study (max. 54 months after FPI)
  Proportion of patients without phlebotomy from treatment start until respective time point
Drug safety | From time of treatment start until end of study (max. 54 months after FPI)
  Incidence of serious adverse events (SAEs), adverse drug reactions (ADRs) and serious adverse drug reactions (SADRs) related to ropeginterferon alfa-2b as characterized by severity, and seriousness
Dosing | From start until end of treatment (max. 54 months after FPI)
  Dose intensity (average dose in µg/4 weeks) and dose over time per patient and overall
Treatment discontinuation | From start until end of treatment (max. 54 months after FPI)
  Frequency of treatment discontinuation and reasons thereof
(S)ADRs leading to permanent treatment discontinuation | From start until end of treatment (max. 54 months after FPI)
  Frequency of patients with (S)ADRs leading to permanent treatment discontinuation
Symptom burden | From time of enrollment until month 36 after treatment start (max. 54 months after FPI)
  Absolute values of single items regarding symptom burden during course of study until month 36.
Treatment reality: previous cytoreductive therapies | From time of treatment start until end of study (max. 54 months after FPI)
  Frequency of distinct previous cytoreductive therapies (if applicable)
Treatment reality: Switch to ropeginterferon alfa-2b | From time of treatment start until end of study (max. 54 months after FPI)
  Reason for switch to ropeginterferon alfa-2b (if applicable) (i.e., frequencies of answers per reasons in the physician´s questionnaire)
Treatment reality: parallel cytoreductive therapies | From time of treatment start until end of study (max. 54 months after FPI)
  Frequency of parallel cytoreductive therapies (combinations)
Treatment reality: subsequent cytoreductive therapies | From time of treatment start until end of study (max. 54 months after FPI)
  Frequency of subsequent cytoreductive therapies (switch to another therapeutic agent)

CONTACTS AND LOCATIONS:
Overall Officials: Eyck von der Heyde, Dr., Principal Investigator — Onkologische Schwerpunktpraxis
Locations (1):
- Onkologisches Studienzentrum Dr. med. Ingo Zander & Dr. med. Eyck von der Heyde, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No